CLINICAL TRIAL: NCT04709731
Title: Cardiovascular Assessment of Ponatinib as Third Line Treatment Option in Chronic Phase Chronic Myeloid Leukemia After Failure of Imatinib and Bosutinib (CarPAs)
Brief Title: Cardiovascular Assessment of Ponatinib as Third Line Treatment in Chronic Phase Chronic Myeloid Leukemia
Acronym: CarPAs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Associazione Italiana Pazienti Leucemia Mieloide Cronica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssociazioneIPLMC; 2018-001334-18 (EudraCT Number)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: Chronic Myeloid Leukemia; Chronic Phase; Ponatinib; BCR-ABL Positive (BCR-ABL+); Philadelphia Chromosome Positive (Ph+); Imatinib and/or Bosutinib Intolerance; Imatinib and/or Bosutinib Resistance
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total Patients (Experimental): Intolerant Group Ponatinib 15 mg tablet, taken orally once daily (QD) Resistant Group Ponatinib 30 mg tablet, taken orally once daily (QD) The dose will be reduced to 15mg once daily (QD) as soon as a Complete Cytogenetic Response will be obtained. In those patients showing Major Molecular Response or better, the dose could be further reduced to 15MG every other day (EOD), due to the prolonged half-life of the drug.
  Interventions: Drug: Ponatinib 15mg QD; Drug: Ponatinib 30mg QD

INTERVENTIONS:
Drug: Ponatinib 15mg QD — Ponatinib 15 mg tablet, taken orally once daily
  Other Names: ICLUSIG; AP24534
Drug: Ponatinib 30mg QD — Ponatinib 30 mg tablet, taken orally once daily
  Other Names: ICLUSIG; AP24534

SUMMARY:
This study will address the therapeutic activity and the safety/biological profile of Ponatinib when used as third line therapy of Chronic Myeloid Leukemia in Chronic Phase after the only two TKIs known for their cardiovascular safety, i.e. Imatinib and Bosutinib.

DETAILED DESCRIPTION:
Phase 2, single-arm, multicentre, open label study which aims to investigate the therapeutic activity and the cardiovascular safety profile of Ponatinib when used as third line therapy of Chronic Myeloid Leukemia in Chronic Phase, after using the only two Tyrosine Kinase Inhibitors (TKIs) known for the safest cardiovascular profile, i.e. Imatinib and Bosutinib. Patients will be stratified according to the cause of discontinuation of the second TKI: intolerance or resistance. The safety of Ponatinib will be assessed by a combination of clinical tests such as ECG, Doppler ultrasound studies to assess arterial and venous vessels, blood pressure monitoring and lipid profiles, combined with inflammatory cytokine analysis which is a known predictor of subsequent cardiovascular adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent approved by Local Ethical Committee before any protocol-specific screening procedures.
2. CML diagnosis, Chronic Phase (CP), treated with imatinib and bosutinib. Previous treatment with dasatinib or nilotinib will not be allowed.
3. Resistant or intolerant to imatinib and/or bosutinib.
4. Able to take oral therapy.
5. Female or male, 18 years of age or older.
6. ECOG performance status 0-2.
7. Minimum life expectancy of 3 months or more.
8. Adequate organ function as defined by the following criteria:

   * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin ≤ 1.5 x ULN (except patients with documented Gilbert's syndrome)
   * Creatinine ≤ 1.5 x ULN
   * Prothrombin time (PT) < 1.5 × ULN
   * Lipase ≤ 1.5 × ULN for institution
   * Amylase ≤ 1.5 × ULN for institution
9. Normal QTcF interval on screening electrocardiogram (ECG) evaluation, defined as QTcF of ≤ 450 ms in males or ≤ 470 ms in females.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
11. Female and male patients who are of childbearing potential must agree to use an effective form of contraception (2 forms of contraception) with their partners throughout participation in this study and for at least 90 days after the last dose of treatment.
12. For females of childbearing potential, a negative pregnancy test must be documented prior to enrolment.

Exclusion Criteria:

1. Current treatment on another therapeutic clinical trial.
2. Received TKI therapy within 7 days prior to receiving the first dose of ponatinib, or have not recovered (> grade 1 by NCI CTCAE, v. 4.0) from AEs (except alopecia) due to agents previously administered.
3. Underwent autologous or allogeneic stem cell transplant < 60 days prior to receiving the first dose of ponatinib; any evidence of on-going graft versus-host disease (GVHD), or GVHD requiring immunosuppressive therapy.
4. Take medications that are known to be associated with Torsades de Pointes.
5. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy.
6. Have previously been treated with ponatinib.
7. Have active central nervous system (CNS) disease as evidenced by cytology or pathology. In the absence of clinical CNS disease, lumbar puncture is not required. History itself of CNS involvement is not exclusionary if CNS has been cleared with a documented negative lumbar puncture.
8. Have significant or active cardiovascular disease, specifically including, but not restricted to:

   1. Myocardial infarction within 3 months prior to first dose of ponatinib,
   2. History of clinically significant atrial arrhythmia or any ventricular arrhythmia,
   3. Unstable angina within 3 months prior to first dose of ponatinib,
   4. Congestive heart failure within 3 months prior to first dose of ponatinib.
9. Have a significant bleeding disorder unrelated to CML or Ph+ ALL.
10. Have a history of pancreatitis or alcohol abuse.
11. Have uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL).
12. Have malabsorption syndrome or other gastrointestinal illness that could affect absorption of orally administered ponatinib.
13. Have been diagnosed with another primary malignancy within the past 3 years (except for non-melanoma skin cancer or cervical cancer in situ, or controlled prostate cancer, which are allowed within 3 years).
14. Pregnancy or breastfeeding.
15. Underwent major surgery (with the exception of minor surgical procedures, such as catheter placement or BM biopsy) within 14 days prior to first dose of ponatinib.
16. Have ongoing or active infection (including known history of human immunodeficiency virus [HIV], hepatitis B virus [HBV], or hepatitis C virus [HCV]). Testing for these viruses is not required in the absence of history.
17. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Exposure adjusted Rate of Arterial Occlusive Events and Serious Arterial Occlusive Events at 1 year after study treatment initiation of each patient | 1 year
  Exposure adjusted Rate of Arterial Occlusive Events (AOE) and Serious AOE (SOE) at 1 year after study treatment initiation of each patient

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gambacorti, Principal Investigator — Ospedale San Gerardo - Monza (MI)
Locations (13):
- Italy (13):
  - Presidio Ospedaliero "Oncologico Businco" - Cagliari (CA), Cagliari
  - AOU "Policlinico Vittorio Emanuele" - Catania (CT), Catania
  - Ospedale San Gerardo - Monza (MB), Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Milano (MI), Milan
  - Azienda Ospedaliera Universitaria "Federico II" - Napoli (NA), Napoli
  - Fondazione IRCCS Policlinico San Matteo - Pavia (PV), Pavia
  - Grande Ospedale Metropolitano "Bianchi-Melacrino-Morelli" - Reggio Calabria (RC), Reggio Calabria
  - AUSL Reggio Emilia (RE), Reggio Emilia
  - ASL Roma 2 "Ospedale S. Eugenio" - Roma (RM), Roma
  - AOU Policlinico Umberto I "Università La Sapienza" - Roma (RM), Roma
  - Azienda Ospedaliero-Universitaria Senese - Siena (SI), Siena
  - AOU Città della Salute e della Scienza - Torino (TO), Torino
  - AOU Integrata Verona "Ospedale Borgo Roma" - Verona (VN), Verona

IPD SHARING:
Plan to Share IPD: No